CLINICAL TRIAL: NCT06005935
Title: Sex-Specific Environmental and Reproductive Health Risk Factors for Lewy Body Dementia
Brief Title: Environmental and Reproductive Health Risk for Lewy Body Dementia
Acronym: LBD-TOROS
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: The Lewy Body Dementia Association (LBDA) (Unknown)
Responsible Party: Principal Investigator, Ece Bayram, Principal Investigator, University of California, San Diego
Other Study IDs: 805745
Record Dates: First submitted 2023-08-15; First posted 2023-08-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Lewy Body Dementia; Parkinson Disease Dementia; Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Lewy body dementia: 50 women and 50 men with a clinical diagnosis of Lewy body dementia (Parkinson's disease dementia or dementia with Lewy bodies) will be included. If assistance is needed to complete the survey, care partners can help, however, they cannot answer the questions on the participant's behalf without the participant's contribution.
  Interventions: Other: Survey
- Controls: 50 women and 50 men with normal cognition and without Parkinson's disease will be included. Normal cognition will be determined using a screening questionnaire in the beginning of the survey to determine eligibility.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Participants will complete a one-time survey including questions on demographics, health status, reproductive health history, environmental and occupational factors one may or may not have been exposed to. The survey can be completed online or over the phone, and should last approximately 30-45 minutes.

SUMMARY:
The goal of this survey study is to identify environmental, occupational and reproductive health risk factors for Lewy body dementia, which includes Parkinson's disease dementia and dementia with Lewy bodies. Participants will complete a one-time survey online or over the phone that includes questions on environmental, occupational factors they may have been exposed to and on medical history including reproductive health. Researchers will then compare the responses of people with Lewy body dementia and people without Parkinson's or memory/thinking problems to see which factors play a role in Lewy body dementia. Identifying risk factors can guide future treatment efforts and provide more insight to this dementia.

DETAILED DESCRIPTION:
Lewy body dementia, including Parkinson's disease dementia and dementia with Lewy bodies, is one of the most common dementias and does not have a cure for now. It can occur differently for women and men, although we are not sure why. The ratio of women to men for the disease prevalence changes with older age, suggesting a potential role for reproductive factors, particularly for women. Environmental factors impact the risk for other types of dementia, although such factors have not been clearly described in Lewy body dementia specifically. Women and men may get exposed to different environmental and occupational risk factors, and the impact of factors can differ for women and men. By using one-time survey that can be completed online or over the phone, we will try to understand which environmental, occupational or reproductive health factors play a role in Lewy body dementia for women and men. By comparing the survey responses of people with Lewy body dementia and people without Parkinson's or memory/thinking problems, we aim to identify specific risk factors for women and men that can guide future treatment efforts and provide more insight into this dementia.

ELIGIBILITY:
Inclusion Criteria:

* For participants with Lewy body dementia: Clinical diagnosis of Lewy body dementia (Parkinson's disease dementia or dementia with Lewy bodies)
* For controls: Normal cognition
* Implication of consent to participate by stating consent verbally over the phone or by selecting the appropriate response on the online survey to indicate consent

Exclusion Criteria:

* For controls: Parkinson's disease or dementia diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with Lewy body dementia will include 50 women and 50 men with a clinical diagnosis of Lewy body dementia (Parkinson's disease dementia or dementia with Lewy bodies). If assistance is needed to complete the survey, care partners can help, however, they cannot answer the questions on the participant's behalf without the participant's contribution. Controls will include 50 women and 50 men with similar age as the participants with Lewy body dementia. Normal cognition will be determined using a screening questionnaire in the beginning of the survey to determine eligibility.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Environmental, occupational, reproductive health factors | 1 year
  Responses of participants with Lewy body dementia and controls completing the survey including questions on environmental, occupational and reproductive health factors will be compared to determine which factors play a role in Lewy body dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Bayram, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information on the study — https://www.lbda.org/men-are-at-greater-risk-for-lewy-body-dementia-than-women-but-why-new-study-seeks-answers/